CLINICAL TRIAL: NCT03051516
Title: HPV Vaccine to Interrupt Progression of Vulvar and Anal Neoplasia (VIVA) Trial: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: HPV Vaccine Therapy in Interrupting Progression in Patients With High-Grade Vulvar or Anal Lesions
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated early due to futility.
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Margaret M. Madeleine, PhD, Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 9790; NCI-2017-00151 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9790 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA213130 (NIH); RG1001522 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: High Grade Anal Canal Intraepithelial Neoplasia; High Grade Vulvar Squamous Intraepithelial Lesion
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (recombinant human papillomavirus nonavalent vaccine) (Experimental): Patients receive recombinant human papillomavirus nonavalent vaccine IM at baseline, 2 months, and 6 months.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration; Biological: Recombinant Human Papillomavirus Nonavalent Vaccine
- Arm II (placebo) (Placebo Comparator): Patients receive placebo IM at baseline, 2 months, and 6 months.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Given IM
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies
Biological: Recombinant Human Papillomavirus Nonavalent Vaccine — Given IM
  Other Names: Gardasil 9; Nonavalent HPV Vaccine; Recombinant HPV Nonavalent Vaccine; Recombinant Human Papillomavirus 9-valent Vaccine
  Arms: Arm I (recombinant human papillomavirus nonavalent vaccine)

SUMMARY:
This phase IV trial studies how well human papillomavirus (HPV) vaccine therapy works in interrupting progression in patients with high-grade vulvar or anal lesions. Vaccines made from HPV peptides or antigens may help the body build an effective immune response to kill tumor cells and decrease the chance of vulvar or anal lesions to progress or come back.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive recombinant human papillomavirus nonavalent vaccine intramuscularly (IM) at baseline, 2 months, and 6 months.

ARM II: Patients receive placebo IM at baseline, 2 months, and 6 months.

After completion of study treatment, patients are followed up at months 7, 12, 18, 24, 36, and 42.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of initial or recurrent anal or vulvar high-grade squamous intraepithelial lesion (AIN2/3 or VIN2/3) diagnosed on or after 1/1/2014; study pathologist will use p16 staining as needed to rule out low-grade squamous intraepithelial lesion (LSIL) disease
* >= 2 months since last therapy for HSIL
* No clinical evidence of HSIL on screening examination; if HSIL is suspected, a biopsy will be done to exclude HSIL; patients whose screening visit reveals HSIL on biopsy, may be re-screened >= 2 months after therapy
* Resident in the catchment area of the clinics and willing to attend up to 8 clinic visits for a 36-month period
* Sexually active women of child-bearing potential must be willing to use effective contraception through month 7 of the study
* If human immunodeficiency virus (HIV) positive, receipt of anti-retroviral therapy continuously for at least 6 months prior to enrollment
* Ability to give informed consent
* Willingness to sign medical records release form and tissue release form

Exclusion Criteria:

* Currently pregnant
* Chemotherapy (current, within the last month, or anticipated in the next 7 months)
* Prior history of invasive HPV-related anogenital cancer (cervical, vaginal, vulvar, penile, or anal cancer), or oropharyngeal cancer (base of tongue, tonsil); prior cancer at other sites (including most of oral cavity) or larynx are not exclusions
* Unstable medical condition (e.g., another malignancy requiring treatment, malignant hypertension, poorly controlled diabetes, another cancer except for fully excised non-melanoma skin cancer)
* Prior HPV vaccination
* Known allergy or intolerance to lidocaine
* Currently participating in an interventional research study related to HPV, except the Anal Cancer HSIL Outcomes Research (ANCHOR) study (NCT02135419)
* Any other condition which, in the opinion of the investigator, may compromise the subject's ability to follow study procedures and safely complete the study

Ages: 27 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Wald, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (2):
- United States (2):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stankiewicz Karita HC, Hauge K, Magaret A, Mao C, Schouten J, Grieco V, Xi LF, Galloway DA, Madeleine MM, Wald A. Effect of Human Papillomavirus Vaccine to Interrupt Recurrence of Vulvar and Anal Neoplasia (VIVA): A Trial Protocol. JAMA Netw Open. 2019 Apr 5;2(4):e190819. doi: 10.1001/jamanetworkopen.2019.0819. PMID 30977845

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment was open between August 2017 and December 2021. Potential participants were recruited through the Fred Hutchinson Cancer Surveillance System and referral by local healthcare providers. Screening took place via phone interviews and in-person visits at the study clinics. Enrollment took place at the two study clinics: Virology Research Center at the University of Washington, and the Center for Women's Reproductive Health at the University of Alabama Birmingham.
Period: Overall Study
Arm/Group | Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) | Arm II (Placebo)
Started | 93 | 95
Vaccination 1 | 93 | 95
Vaccination 2 | 91 | 94
Vaccination 3 | 83 | 90
Month 7 Follow-Up | 80 | 87
Month 12 Follow-Up | 78 | 81
Month 18 Follow-Up | 66 | 75
Month 24 Follow-Up | 59 | 70
Month 36 Follow-Up | 44 | 53
Completed | 38 | 42
Not Completed | 55 | 53

BASELINE CHARACTERISTICS:
Population: Participants who have completed Enrollment Visit and had at least 30 days follow-up after the initial dose of vaccine (n=185) were included in the intention-to-treat analysis and are considered part of the Baseline Analysis Population. Three participants (2 in Arm I/vaccine and 1 in Arm II/placebo) were excluded from analysis due to completing only one vaccination before study exit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) | Arm II (Placebo) | Total
Number analyzed (Participants) | 91 | 94 | 185
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [47 to 61] | 57 [51 to 63] | 55 [48 to 62]
Sex/Gender, Customized [Number; unit: participants]
  Women | 49 | 50 | 99
  Men | 41 | 44 | 85
  Transgender women | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 3 | 8
  Not Hispanic or Latino | 84 | 89 | 173
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 6 | 15
  White | 70 | 75 | 145
  More than one race | 5 | 7 | 12
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 91 | 94 | 185
Anatomic Site of HSIL (high-grade squamous intraepithelial lesion) [Count of Participants; unit: Participants]
  Anal | 50 | 53 | 103
  Vulvar | 41 | 41 | 82
Smoking Status [Count of Participants; unit: Participants]
  Never | 40 | 52 | 92
  Former | 31 | 24 | 55
  Current | 20 | 18 | 38
HIV Status [Count of Participants; unit: Participants]
  HIV Positive | 32 | 39 | 71
  HIV Negative | 59 | 55 | 114

OUTCOME MEASURES:

1. Primary Outcome: Persistent High-risk Infection Among Vaccine Compared With Placebo Recipients
Description: Persistence will be measured as two or more consecutive polymerase chain reaction (PCR) positive swabs for the same human papillomavirus (HPV) genotype. Will use Chi-Square test to compare the number of participants with the persistent infection in the vaccinated to unvaccinated group.
Time Frame: Up to month 36
Population: Participants were included in this analysis if they had 2 or more HPV DNA PCR results from swabs collected after the baseline swab. Of the 185 participants in the baseline population, 117 were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 53 | 64
Participants
  HPV16 persistence identified | 7 | 9
  HPV18/45 persistence identified | 3 | 5
  HPV31/33/52/58 persistence identified | 3 | 11
  HPV33/39/51/56/59 persistence identified | 4 | 8
  Overall high-risk HPV persistence identified | 13 | 21
  High-risk HPV persistence NOT identified | 23 | 10
Statistical Analysis 1: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); This p-value compares HPV16 persistence by study arm; Test type: Superiority; p = 0.89, Chi-squared
Statistical Analysis 2: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); This p-value compares HPV18/45 persistence by study arm; Test type: Superiority; p = 0.65, Chi-squared
Statistical Analysis 3: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); This p-value compares HPV31/33/52/58 persistence by study arm; Test type: Superiority; p = 0.056, Chi-squared
Statistical Analysis 4: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); This p-value compares HPV35/39/51/56/59 persistence by study arm; Test type: Superiority; p = 0.38, Chi-squared
Statistical Analysis 5: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); Test type: Superiority; p = 0.33, Chi-squared — This p-value compares overall HPV persistence and is not specific to HPV genotype

2. Secondary Outcome: Time to Recurrence of Anogenital High Grade Squamous Intraepithelial Lesion (HSIL)
Description: Will compare vaccine and placebo recipients. Will evaluate differences in the hazard of recurrence using Cox proportional hazards in the intention to treat population and the per protocol population.
Time Frame: Up to month 36
Measure: Number; unit: Recurrent events per 100 person-years
Arm/Group | Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 91 | 94
Recurrent events per 100 person-years | 8.1 | 10.1
Statistical Analysis 1: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); Test type: Superiority; p = 0.54, Log Rank

3. Secondary Outcome: Incidence of Adverse Events (AEs) Via Solicited Vaccine Reactogenicity by Arm
Description: Will monitor safety by comparing type and frequency of AEs in the two study arms, graded according to the Food and Drug Administration criteria. Symptoms are reported at least once from any dose.
Time Frame: Up to month 36
Population: There were 173 incidence of reported symptoms among participants in Arm I (Vaccine) and 127 incidence of reported symptoms among participants in Arm II (Placebo). Overall, there were 91 participants in Arm I (Vaccine) and 94 participants in Arm II (Placebo) reported symptoms at least once for any dose received.
Measure: Count of Units; unit: Symptom reports
Units Other Than Participants: Symptom reports
Arm/Group | Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 91 | 94
Number analyzed (Symptom reports) | 173 | 127
Symptom reports
  Fever or chills | 6 | 2
  Headache | 24 | 22
  Fatigue | 23 | 25
  Muscle aches | 17 | 17
  Pain at injection site | 33 | 17
  Tenderness at injection site | 53 | 31
  Swelling at injection site | 12 | 2
  Medical attention/medication | 5 | 11
Statistical Analysis 1: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); This comparison is specific to the incidence of fever or chills; Test type: Other — Descriptive analysis; p = 0.135, Chi-squared
Statistical Analysis 2: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); This comparison is specific to the incidence of headache; Test type: Other — Descriptive analysis; p = 0.640, Chi-squared
Statistical Analysis 3: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); This comparison is specific to the incidence of fatigue; Test type: Other — Descriptive analysis; p = 0.838, Chi-squared
Statistical Analysis 4: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); This comparison is specific to the incidence of muscle aches; Test type: Other — Descriptive analysis; p = 0.917, Chi-squared
Statistical Analysis 5: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); This comparison is specific to the incidence of pain at injection site; Test type: Other — Descriptive analysis; p = 0.005, Chi-squared
Statistical Analysis 6: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); This comparison is specific to the incidence of tenderness at injection site; Test type: Other — Descriptive analysis; p = 0.001, Chi-squared
Statistical Analysis 7: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); This comparison is specific to the incidence of swelling at injection site; Test type: Other — Descriptive analysis; p = 0.004, Chi-squared
Statistical Analysis 8: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) vs Arm II (Placebo); This comparison is specific to the incidence of medical attention/medication required; Test type: Other — Descriptive analysis; p = 0.133, Chi-squared

4. Secondary Outcome: HPV Antibody Level
Description: Will evaluate placebo and vaccine recipients separately. Will assess whether presence and amount of HPV antibody, detected at baseline in the placebo arm, is protective against recurrence. For the vaccine arm, will assess whether magnitude of vaccine antibody levels month 1 following the third vaccination in the vaccine arm affects recurrence.
Time Frame: Up to month 36
Population: Participants with usable serology samples from at least one timepoint are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) | Arm II (Placebo)
Number analyzed (Participants) | 68 | 80
Participants
  HPV16: Negative, No event | 33 | 49
  HPV16: Positive, no event | 22 | 13
  HPV16: Negative, HSIL | 8 | 12
  HPV16: Positive, HSIL | 5 | 6
  HPV18: Negative, No event | 32 | 48
  HPV18: Positive, no event | 23 | 14
  HPV18: Negative, HSIL | 7 | 12
  HPV18: Positive, HSIL | 6 | 6
  HPV31: Negative, No event | 28 | 48
  HPV31: Positive, no event | 27 | 14
  HPV31: Negative, HSIL | 8 | 13
  HPV31: Positive, HSIL | 5 | 5
  HPV33: Negative, No event | 30 | 47
  HPV33: Positive, no event | 25 | 15
  HPV33: Negative, HSIL | 8 | 15
  HPV33: Positive, HSIL | 5 | 3
  HPV45: Negative, No event | 33 | 41
  HPV45: Positive, no event | 22 | 21
  HPV45: Negative, HSIL | 8 | 16
  HPV45: Positive, HSIL | 5 | 2
  HPV52: Negative, No event | 27 | 42
  HPV52: Positive, no event | 28 | 20
  HPV52: Negative, HSIL | 7 | 14
  HPV52: Positive, HSIL | 6 | 4
  HPV58: Negative, No event | 28 | 44
  HPV58: Positive, no event | 27 | 18
  HPV58: Negative, HSIL | 7 | 13
  HPV58: Positive, HSIL | 6 | 5
  Any HPV: Negative, No event | 16 | 20
  Any HPV: Positive, no event | 39 | 42
  Any HPV: Negative, HSIL | 4 | 6
  Any HPV: Positive, HSIL | 9 | 12
Statistical Analysis 1: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine); This p-value compares HSIL recurrence and presence of HPV16, in Arm I (Vaccine); Test type: Superiority; p = 0.93, Log Rank
Statistical Analysis 2: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine); This p-value compares HSIL recurrence and presence of HPV18, in Arm I (Vaccine); Test type: Superiority; p = 0.77, Log Rank
Statistical Analysis 3: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine); This p-value compares HSIL recurrence and presence of HPV31, in Arm I (Vaccine); Test type: Superiority; p = 0.57, Log Rank
Statistical Analysis 4: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine); This p-value compares HSIL recurrence and presence of HPV33, in Arm I (Vaccine); Test type: Superiority; p = 0.73, Log Rank
Statistical Analysis 5: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine); This p-value compares HSIL recurrence and presence of HPV45, in Arm I (Vaccine); Test type: Superiority; p = 0.998, Log Rank
Statistical Analysis 6: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine); This p-value compares HSIL recurrence and presence of HPV52, in Arm I (Vaccine); Test type: Superiority; p = 0.93, Log Rank
Statistical Analysis 7: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine); This p-value compares HSIL recurrence and presence of HPV58, in Arm I (Vaccine); Test type: Superiority; p = 0.95, Log Rank
Statistical Analysis 8: Comparison: Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine); This p-value compares HSIL recurrence and presence of any HPV type, in Arm I (Vaccine); Test type: Superiority; p = 0.91, Log Rank
Statistical Analysis 9: Comparison: Arm II (Placebo); This p-value compares HSIL recurrence and presence of HPV16, in Arm II (Placebo); Test type: Superiority; p = 0.22, Log Rank
Statistical Analysis 10: Comparison: Arm II (Placebo); This p-value compares HSIL recurrence and presence of HPV18, in Arm II (Placebo); Test type: Superiority; p = 0.27, Log Rank
Statistical Analysis 11: Comparison: Arm II (Placebo); This p-value compares HSIL recurrence and presence of HPV31, in Arm II (Placebo); Test type: Superiority; p = 0.72, Log Rank
Statistical Analysis 12: Comparison: Arm II (Placebo); This p-value compares HSIL recurrence and presence of HPV33, in Arm II (Placebo); Test type: Superiority; p = 0.71, Log Rank
Statistical Analysis 13: Comparison: Arm II (Placebo); This p-value compares HSIL recurrence and presence of HPV45, in Arm II (Placebo); Test type: Superiority; p = 0.11, Log Rank
Statistical Analysis 14: Comparison: Arm II (Placebo); This p-value compares HSIL recurrence and presence of HPV52, in Arm II (Placebo); Test type: Superiority; p = 0.58, Log Rank
Statistical Analysis 15: Comparison: Arm II (Placebo); This p-value compares HSIL recurrence and presence of HPV58, in Arm II (Placebo); Test type: Superiority; p = 0.81, Log Rank
Statistical Analysis 16: Comparison: Arm II (Placebo); This p-value compares HSIL recurrence and presence of any HPV type, in Arm II (Placebo); Test type: Superiority; p = 0.73, Log Rank

ADVERSE EVENTS:
Time Frame: 42 months, from enrollment visit (Month 0) to final follow-up at Month 42.
Arm/Group | Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 5/91 | 2/94
Serious Adverse Events (participants affected / at risk) | 19/91 | 16/94
Other Adverse Events (participants affected / at risk) | 60/91 | 58/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) (N=91) | Arm II (Placebo) (N=94)
Fracture, right femur (Injury, poisoning and procedural complications) | 1 | 0
Fracture, right hip (Injury, poisoning and procedural complications) | 1 | 0
Fracture, right arm (Injury, poisoning and procedural complications) | 1 | 0
Fracture, left leg (Injury, poisoning and procedural complications) | 1 | 0
Fracture, broken neck (Injury, poisoning and procedural complications) | 1 | 0
Hospitalization due to multiple abscesses (Infections and infestations) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Small bowel obstruction (Gastrointestinal disorders) | 0 | 1
Pyelonephritis (Renal and urinary disorders) | 0 | 1
Probable gastroenteritis, 3-day hospitalization (Gastrointestinal disorders) | 0 | 1
COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Severe migraine requiring overnight hospitalization (General disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Death due to COVID-19 related complications (Infections and infestations) | 0 | 1
Invasive lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
High grade locally advanced squamous cell carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Angina (Cardiac disorders) | 0 | 1
Skin Infection, left arm (Infections and infestations) | 0 | 1
Deceased due to unknown cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
deceased, secondary to metastatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Coma secondary to fall (Nervous system disorders) | 1 | 0
Ischemic stroke (Nervous system disorders) | 1 | 0
Severe sepsis from atypical/viral pneumonia (Infections and infestations) | 1 | 0
Pneumonia requiring inpatient hospitalization and intubation (Infections and infestations) | 1 | 0
Pancreatitis or Gatroenteritis (General disorders) | 1 | 0
Skin and soft tissue infection/abscess secondary to Staph aureus (MRSA) (Infections and infestations) | 1 | 0
Alcohol-related pancreatitis (Endocrine disorders) | 1 | 0
Transurethral resections of the prostate (Surgical and medical procedures) | 1 | 0
Inguinal hernia repair with subsequent urinary retention (Surgical and medical procedures) | 1 | 0
Motor vehicle accident (Injury, poisoning and procedural complications) | 1 | 0
Acute pancreatitis (Endocrine disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Recombinant Human Papillomavirus Nonavalent Vaccine) (N=91) | Arm II (Placebo) (N=94)
Knot on left arm post COVID-19 injection (General disorders) | 0 | 1
Sore arm post COVID-19 injection (General disorders) | 0 | 1
Fatigue post COVID-19 injection (General disorders) | 0 | 1
High fever (101-102 degrees) post COVID-19 injection (General disorders) | 0 | 1
Weakness post COVID-19 injection (General disorders) | 0 | 1
Fatigue (General disorders) | 23 | 26
Throbbing in right big toe (General disorders) | 0 | 1
Throbbing in right collar bone (General disorders) | 0 | 1
Spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Fever or chills (Infections and infestations) | 6 | 8
Headache (General disorders) | 24 | 22
Muscle aches (General disorders) | 17 | 17
Injection site pain (Injury, poisoning and procedural complications) | 33 | 17
Injection site tenderness (Injury, poisoning and procedural complications) | 53 | 31
Injection site swelling (Injury, poisoning and procedural complications) | 12 | 2
Medical attention or medication required (General disorders) | 5 | 11

LIMITATIONS AND CAVEATS:
An interim analysis found the intervention to be futile. Therefore, the VIVA trial was ended effective July 31st, 2022, for the University of Washington clinic, and December 31st, 2022, for the University of Alabama Birmingham clinic. Participants were offered the choice of continuing any outstanding visits until the end of the study at the respective sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03051516/Prot_SAP_002.pdf
  • Informed Consent Form (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03051516/ICF_001.pdf